CLINICAL TRIAL: NCT06470555
Title: A Randomised Controlled Trial to Compare Manual Compression and Suture-mediated Haemostasis After Catheter Ablation of Atrial Fibrillation
Brief Title: Haemostasis After Venous Access in Atrial Fibrillation Catheter Ablation: The HARNESS Trial
Acronym: HARNESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRAS 345085
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Atrial Fibrillation; Femoral Vein Injury; Bleeding
Keywords: Atrial fibrillation; Catheter ablation; Femoral haemostasis
MeSH Terms: conditions — Atrial Fibrillation; Hemorrhage

STUDY DESIGN:
Intervention Model Description: Patients will be randomised into one of three strategies for haemostasis (with a final allocation ratio of 1:1:1):
  * Conventional arm: Manual compression with 4-hours of bed rest;
  * Intervention arm 1: A figure-of-eight suture secured with a three-way tap (Fo8s-3wt) with 4-hours of bed rest;
  * Intervention arm 2: A Fo8s-3wt with 2-hours of bed rest.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Manual compression with 4-hours of bed rest (Active Comparator): Femoral haemostasis using manual compression. Bed rest duration of 4 hours following initial haemostasis.
  Interventions: Other: Manual compression; Other: Conventional bed rest duration of 4-hours
- A figure-of-eight suture secured with a three-way tap with 4-hours of bed rest; (Experimental): Femoral haemostasis using a figure-of-eight suture secured with a three-way tap.
  Bed rest duration of 4 hours following initial haemostasis.
  Interventions: Other: A figure-of-eight suture secured with a three-way tap; Other: Conventional bed rest duration of 4-hours
- A figure-of-eight suture secured with a three-way tap with 2-hours of bed rest; (Experimental): Femoral haemostasis using a figure-of-eight suture secured with a three-way tap.
  Bed rest duration of 2 hours following initial haemostasis.
  Interventions: Other: A figure-of-eight suture secured with a three-way tap; Other: Shortened bed rest duration of 2-hours

INTERVENTIONS:
Other: A figure-of-eight suture secured with a three-way tap — Femoral haemostasis using a figure-of-eight suture technique
  Arms: A figure-of-eight suture secured with a three-way tap with 2-hours of bed rest;; A figure-of-eight suture secured with a three-way tap with 4-hours of bed rest;
Other: Shortened bed rest duration of 2-hours — Bed rest duration of 2-hours after initial haemostasis
  Arms: A figure-of-eight suture secured with a three-way tap with 2-hours of bed rest;
Other: Manual compression — Femoral haemostasis using manual compression
  Arms: Manual compression with 4-hours of bed rest
Other: Conventional bed rest duration of 4-hours — Bed rest duration of 4-hours after initial haemostasis
  Arms: A figure-of-eight suture secured with a three-way tap with 4-hours of bed rest;; Manual compression with 4-hours of bed rest

SUMMARY:
Atrial fibrillation (AF) is the most common heart rhythm disorder affecting adults in the United Kingdom. In patients with AF who continue to experience symptoms despite medications, catheter ablation is an established interventional treatment. Ablation is performed by inserting a number of plastic tubes in the veins in the groin, in order to access the heart.

Despite continued advances in equipment and techniques, groin complications remain the most common complications after AF ablation. The severity of these can range from minor (e.g. bleeding resolvable with manual pressure) to major (bleeding requiring blood transfusion, prolonged hospitalisation, intervention, or rarely resulting in death).

Following ablation, the plastic tubes in the groin are removed before leaving the procedure room. Once removed, the doctor will stop the bleeding in the groin. There are two commons ways in which the doctor can stop the bleeding: 1) conventional treatment with manual compression - the doctor applies pressure with their hands to the groin area to stop the bleeding; 2) suture treatment (also known as a "stitch") - the doctor inserts a suture to the groin area and secures this in place with a small plastic device (called a three-way tap). The suture and three-way tap are left in place for a few hours before being removed. Both of these methods are commonly in use. However, there is no high-quality evidence to support whether one way is better than the other.

After stopping the bleeding, patients are generally asked to lay flat for 4 hours to prevent any bleeding. It is not known whether this duration can safely be shortened.

The Haemostasis AfteR veNous accESS in AF catheter ablation (HARNESS) trial is a pragmatic, single-centre, open label, randomised controlled trial which will compare a suture with a three-way tap to manual compression, and examine the impact of bed rest duration on clinical outcomes.

ELIGIBILITY:
The trial aims to recruit patients presenting to our institution for AF catheter ablation. Potential participants will be assessed against a two-tiered set of inclusion and exclusion criteria.

Inclusion Criteria for Pre-Lab Phase - Screening and Consent:

Patients scheduled for AF catheter ablation with proposed femoral venous access, regardless of their gender identity, ethnicity and religious belief.

Exclusion Criteria for Pre-Lab Phase - Screening and Consent:

* ≤ 18 years of age
* Planned bilateral femoral venous access
* Planned femoral arterial access
* Any haematoma at planned puncture site prior to femoral sheath insertion
* Established diagnosis of any haematologic disorder or genetic defect predisposing to bleeding
* Inability to perform adequate consent:

  * Communication issues (e.g. mental capacity, forgotten glasses)
  * Inadequate time for the participant to read and consider trial
  * Unscheduled Urgent or Emergency procedures
* Patients who are scheduled to be transferred to other hospitals ("treat and return") before haemostasis is achieved.
* Electronic patient record technical failure leading to an inability to record participants' care

Inclusion Criteria for In-Lab Phase - Before Randomisation

Four or fewer femoral venous sheaths in situ (size range: 6 Fr to 17 Fr) with planned removal in lab

Exclusion Criteria for In-lab Phase - Before Randomisation

* Sizeable (>5cm) puncture-related haematoma requiring manual compression prior to femoral venous sheath removal
* Presence of femoral arterial sheath
* Clinically suspected femoral arterial puncture
* Patient leaving lab with femoral venous sheath in situ
* Randomisation system not available
* A change in patient's clinical condition during procedure deemed by the operator sufficient to exclude from the trial
* Procedural complication requiring procedure termination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2024-08-27 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
The rate of any femoral venous access site complication from the time of initial haemostasis in the cath lab to end of follow-up. | Patients will be followed up to hospital discharge or to 24 hours after randomisation (whichever is the sooner).
  Defined as:
  1. Bleeding (with or without haematoma formation) at the site of femoral venous access site after initial haemostasis:
     * Grade 1 - overt but minor bleeding requiring minimal bedside action(s) such as manual compression
     * Grade 2 - continuous or significant overt bleeding requiring timely investigation and/or action, such as ultrasound, non-invasive radiological assessment, fluid resuscitation, or blood transfusion
     * Grade 3 - continuous or significant overt bleeding requiring urgent or emergency interventional procedure (interventional radiology or surgical intervention), or resulting in critical illness
     * Grade 4 - continuous or significant overt bleeding resulting in death
     Trial definition of haematoma:
     * Grade 1 - Raised haematoma < 6 cm in longest dimension
     * Grade 2 - Raised haematoma ≥ 6 cm in longest dimension
  2. Development of local subcutaneous infection at the femoral venous access site.

SECONDARY OUTCOMES:
Time from femoral sheath removal to leaving the cath lab | Patients will be followed up to hospital discharge or to 24 hours after randomisation (whichever is the sooner).
  Time (in minutes) from removal of femoral sheath(s) to exiting the cardiac catheter laboratory.
Time from sheath removal to successful mobilisation without femoral venous access site complication | Patients will be followed up to hospital discharge or to 24 hours after randomisation (whichever is the sooner).
  Time (in minutes) from removal of femoral sheath(s) to mobilisation without femoral access site complication.
Time from sheath removal to hospital discharge | Patients will be followed up to hospital discharge or to 24 hours after randomisation (whichever is the sooner).
  Time (in minutes) from removal of femoral sheath(s) to hospital discharge.
Rate of delayed discharge due to the need for femoral venous access site care | Patients will be followed up to hospital discharge or to 24 hours after randomisation (whichever is the sooner).
  Incidence of delayed discharge due to the need for femoral venous access site care.

CONTACTS AND LOCATIONS:
Overall Officials: Dhiraj Gupta, MD, Study Chair — Liverpool Heart and Chest Hospital
Locations (1):
- Liverpool Heart and Chest Hospital Foundation Trust, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No